## Statistical Analysis

The percentage (%) success (0-100%) for each item on each variable was calculated for scores obtained in the FAB and in the performance of the feeding task. The closer to 100, the higher the success rate for each item. For the analysis of the feeding task data, the duration of the following steps was determined: "start the movement" (sec), "grasp the cutlery" (sec), "put food in the cutlery" (sec), "take the cutlery in the mouth "(sec)," put food in the mouth "(sec), were normalized in relation to the total task time (sec). The closer to 100, the higher the success rate for each stage.

Descriptive measures (means and standard deviation) were used to characterize the implementation of READY2E.AT protocol. For the variables: Unilateral Reach training score, Errors in Unilateral Reach training, Reach training score with Memory tasks, Errors in Reach with Memory Tasks, Fine Motricity Training Score, Fine Motricity Training Errors, Motor Reach Sequence Score, Motor Sequence Reach Training Errors, and Total Training Time (minutes).

In order to investigate the existence of significant differences in percentage of success of FAB scores and in feeding performance in the different groups (Group 1 and Group 2), at different times (T0, T1 and T1-T0), non-parametric test for independent samples were implemented.